CLINICAL TRIAL: NCT00704496
Title: The Effect of Pseudoephedrine on Rhinitis and Sleep
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Timothy Craig, Timothy Craig, D.O., Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 25325
Record Dates: First submitted 2008-06-24; First posted 2008-06-25 (Estimated); Results first posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-09

CONDITIONS: Rhinitis; Sleep
Keywords: Sleep, Pseudoephedrine
MeSH Terms: conditions — Rhinitis | interventions — Pseudoephedrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Pseudoephedrine
- Pseudoephedrine (Active Comparator): Pseudoephedrine is a 240 mg PO per day
  Interventions: Drug: Pseudoephedrine

INTERVENTIONS:
Drug: Pseudoephedrine — Pseudoephedrine is a 240 mg PO per day
  Other Names: Placebo

SUMMARY:
The hypothesis is that pseudoephedrine, a sympathomimetic amine commonly used as a decongestant, will decrease nasal congestion leading to increased patency of the nose and a decrease in nighttime sleep fragmentation in individuals with year round perennial allergic rhinitis (PAR). This decrease in sleep fragmentation will reduce daytime somnolence and fatigue.

DETAILED DESCRIPTION:
The hypothesis is that pseudoephedrine, a sympathomimetic amine commonly used as a decongestant, will decrease nasal congestion leading to increased patency of the nose and a decrease in nighttime sleep fragmentation in individuals with year round perennial allergic rhinitis (PAR). This decrease in sleep fragmentation will reduce daytime somnolence and fatigue. We studied patients treated with placebo compared to FDA approved dose of pseudoephedrine and assessed sleep, QOL and daytime sleepiness.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65.
2. History of allergic rhinitis.
3. The ability to be placed on placebo without significant compromise in the quality of life.
4. General good health.
5. Ability to comply with the protocol and sign an informed consent.
6. Have daytime sleepiness by history.
7. Have poor sleep by history.
8. Have fatigue by history.
9. Have a skin test or RAST test to a perennial allergen (indoor mold, dog, cat, mite) with correlating symptoms.

Exclusion Criteria:

1. Age fewer than 18 or over 65 years.
2. A history of sleep apnea.
3. Atopic diseases other than allergic rhinitis, such as atopic dermatitis or asthma.
4. Non-allergic rhinitis.
5. Hypertension
6. Diabetes Mellitus
7. Inability to tolerate pseudoephedrine
8. Significant other diseases as determined by the investigator.
9. Use of a research medication within 30 days.
10. Use of a nasal steroid or topical antihistamine or decongestant within 30 days.
11. Use of beta-blockers, antidepressants, oral decongestants, oral steroids, or H2-blockers.
12. Excessive use of alcohol or drug abuse.
13. Inability to stop medication use during run-in period.
14. Use of an oral antihistamine within 1 week of enrollment.
15. Failed to have benefit when pseudoephedrine was used for rhinitis or asthma in the past

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Craig, D.O., Principal Investigator — Penn State University
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: data disposed of and no longer in existence
Groups:
- Placebo: Placebo arm
Period: Overall Study
Arm/Group | Pseudoephedrine | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: data disposed of and no longer in existence
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pseudoephedrine | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Improvement of Sleep Associated With the Use of Pseudoephedrine as Compared to the Placebo
Description: sleep improvement by subjective questionnaires
Time Frame: 3 years
Population: data disposed of and no longer in existence
Arm/Group | Placebo | Pseudoephedrine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Improvement of Daytime Somnolence With Pseudoephedrine as Compared to Placebo
Description: daytime sleepiness by subjective questionnaires
Time Frame: 3 years
Population: data disposed of and no longer in existence
Arm/Group | Placebo | Pseudoephedrine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Pseudoephedrine
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
data disposed of and no longer in existence

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes